CLINICAL TRIAL: NCT00047853
Title: fMRI Investigation of Explicit Cue and Contextual Fear
Brief Title: Brain Imaging Changes in Fear and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 020321; 02-M-0321
Record Dates: First submitted 2002-10-22; First posted 2002-10-23 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2022-08-02

CONDITIONS: Anxiety Disorders; Fear
Keywords: Stress; Fear; Anxiety; Neuroimaging; Unpredictability; Healthy Volunteer (HV)
MeSH Terms: conditions — Anxiety Disorders | interventions — Reflex, Startle

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Healthy Volunteer (Experimental): Healthy volunteer will undergo Functional magnetic resonance imaging (fMRI) and/or magneto-encephalography (MEG) and will be scanned during runs of either shock or no shock.
  Interventions: Device: Shock device; Device: Acoustic startle
- Patient (Experimental): Participant with a current diagnosis of generalized anxiety disorder (GAD), panic disorder, social anxiety disorder (SAD), specific phobia, posttraumatic stress disorder (PTSD), or major depression will undergo Functional magnetic resonance imaging (fMRI) and will be scanned during runs of either shock or no shock.
  Interventions: Device: Shock device

INTERVENTIONS:
Device: Shock device — A participant could receive a shock or not receive as shock
Device: Acoustic startle — Acoustic startle for MEG only
  Arms: Healthy Volunteer

SUMMARY:
The purpose of this study is to use brain imaging technology to investigate brain changes in people exposed to predictable versus unpredictable unpleasant stimuli. Unpleasant events that can be predicted evoke a response of fear, whereas unpredictable, unpleasant stimuli cause chronic anxiety not associated with a specific event. Information gained from this study may help in the development of more effective treatments for anxiety disorders.

When confronted with fearful events, people eventually develop fear of specific cues that were associated with these events as well as to the environmental context in which the fearful event occurred. Evidence suggests that cued fear and contextual fear model different aspects of anxiety. However, studies that examine the way the brain affects expression of contextual fear have not been conducted. This study will use magnetic resonance imaging (MRI) or Magneto-encephalography (MEG) to compare the brain activity underlying fear brought on by predictable and unpredictable aversive stimuli.

DETAILED DESCRIPTION:
This protocol examines the neurobiology of fear and anxiety using various approaches. During fear conditioning in which a phasic explicit cue (e.g., a light) is repeatedly associated with an aversive unconditioned stimulus (e.g., a shock), the organism develops fear to the explicit cue as well as to the environmental context in which the experiment took place. Experimental evidence suggests that cued fear and contextual fear model different aspects of anxiety. Studies in patients indicated that contextual fear may model an aspect that is especially relevant to anxiety disorders. However, the neural basis for the expression of contextual fear has not previously been elucidated in human imaging studies. One important determinant of contextual fear is predictability: contextual fear increases when a threat (e.g., electric shock) is unpredictable, as opposed to when the threat is predictable. The aim of this study is to compare the neural substrates underlying fear evoked by predictable versus unpredictable shocks. Animal studies have indicated that conditioned responses to predictably cued threat and to less explicit threat are separate processes mediated by distinct brain structures. Psychophysiological data suggest that the proposed procedure can differentiate between these two responses. Hence, we anticipate that this procedure will allow us to compare brain correlates of these responses in humans. Another objective is to study effects of threat of shock on processing and learning of threat cues in the amygdala, the visual and auditory systems, and motivation/reward systems. This will be investigated by means of event-related magneto-encephalography (MEG) and fMRI measurements using various paradigms. Finally, a last project will examine how pharmacologic manipulation of gamma-aminobutyric acid (GABA) levels with the benzodiazepine alprazolam affects the relationship between GABA concentration (quantified with magnetic resonance spectroscopy, MRS), visual- and auditory-induced gamma oscillations (measured with MEG), and fMRI BOLD response.

ELIGIBILITY:
* INCLUSION CRITERIA:

All screening procedures described in this section are conducted under screening protocol 01-M-0254. Subjects must meet the following inclusion criteria in order to participate in the study:

1. Male or female volunteers ages 18-50 years old.
2. Judged to be in good physical health on the basis of medical history, a clinical MRI scan, and physical examination. Physical exams will be conducted by a National Institute of Mental Health (NIMH) credentialed physician or nurse. Clinical laboratory tests will be ordered based on his/her discretion.
3. Healthy subjects judged to be in good psychiatric health on the basis of the Structured Clinical Interview for DSM-IV-TR. The SCID will be administered by a credentialed NIMH clinician.
4. Able to understand procedures and agree to participate in the study by giving written informed consent.
5. This protocol (02-M-0321) will include patients with a primary diagnosis (under the clinical responsibility of Dr. Daniel Pine) of generalized anxiety disorder, panic disorder, SAD, PTSD, specific phobia, and major depression according to Diagnostic and Statistical Manual (DSM)-IV.
6. Subjects will not be asked to completely stop smoking or drinking coffee during this study because they may experience withdrawal symptoms, which could affect our study results. However, they will be asked to abstain from drinking caffeinated beverage including coffee, tea and caffeinated soft drinks and from smoking for at least 1 hour prior to testing. They will also be instructed not to drink alcohol on the night prior to testing and on the day of testing.
7. Speaks English or Spanish fluently (subjects with Major Depressive Disorder, healthy volunteers)
8. Speaks English fluently (subjects with Anxiety Disorder)

EXCLUSION CRITERIA:

Subjects will be excluded from the study if they meet the following exclusion criteria:

1. Clinically significant organic disease, e.g., cardiovascular disease.
2. Clinically significant abnormalities in physical examination.
3. Any medical condition that increases risk for fMRI (e.g. pacemaker, metallic foreign body in eye).
4. History of any disease, which in the investigators opinion may confound the results of the study, including, but not limited to, history of organic mental disorders, seizure, or mental retardation.
5. Have a current diagnosis of alcohol or substance abuse ACCORDING TO DSM IV CRITERIA
6. Have a lifetime diagnosis of alcohol or substance dependence ACCORDING TO DSM IV CRITERIA.
7. Unless subject is enrolled as a patient, subjects should not have current Axis I psychiatric disorders as identified with the Structured Clinical Interview for DSM-IV, non-patient edition (SCID/NP).
8. If a healthy volunteer, past bipolar depression and any history of psychosis or delusional disorders.
9. If a healthy volunteer, first degree relative with history of psychotic disorder such as schizophrenia or bipolar disorder
10. If a healthy volunteer, psychotropic medication within 4 weeks of scanning
11. Medications that act on the central nervous system (e.g., Lorazepam, Codeine) and thus may interfere with the interpretation of study results. Specific exclusionary drug classes include but are not limited to: (opioid analgesics, DA receptor agonists, anticholinergics, monoamine oxidase (MAO) inhibitors, COMT inhibitors, as well as any illicit substances). In addition, healthy participants may not be on psychotropic medications.
12. Pregnancy, i.e., a positive Beta-human chorionic gonadotropin (HCG) urine test conducted prior to each experiment session.
13. Current or past history of cubital tunnel syndrome or carpal tunnel syndrome for shock studies that use the wrist for placement of electrodes. Cubital tunnel and carpal tunnel syndrome are exclusionary only for diagnosis on same arm as electrodes and are not exclusionary for studies that place shocks on ankles or feet.
14. Reynaud's syndrome for the cold pressor test experiment
15. Color blindness (for the active avoidance task only)

ADDITIONAL EXCLUSION CRITERIA FOR PATIENTS:

Patients who would be unable to comply with study procedures or assessments.

Patients will be excluded if they have a current or past history of any psychotic disorder, bipolar disorder, delirium, dementia, amnestic disorder, cognitive disorder not otherwise specified, any of the pervasive developmental disorders, or mental retardation.

Patients (except PTSD) on psychotropic medications within 2 wees of study visits, or within 6 weeks of study visits for fluoxetine will be excluded.

PTSD patients on psychotropics medication within 2 weeks of study visits will be excluded, with the exception of antidepressants, and benzodiazepines; the preceding two classes of medications will not preclude enrollment for PTSD participants only.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1080 (Actual)
Dates: Start 2002-11-04 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryland Pao, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
.We plan to submit de-identified data to the repository.

REFERENCES:
- [Result] Torrisi S, O'Connell K, Davis A, Reynolds R, Balderston N, Fudge JL, Grillon C, Ernst M. Resting state connectivity of the bed nucleus of the stria terminalis at ultra-high field. Hum Brain Mapp. 2015 Oct;36(10):4076-88. doi: 10.1002/hbm.22899. Epub 2015 Jul 14. PMID 26178381
- [Result] Torrisi S, Nord CL, Balderston NL, Roiser JP, Grillon C, Ernst M. Resting state connectivity of the human habenula at ultra-high field. Neuroimage. 2017 Feb 15;147:872-879. doi: 10.1016/j.neuroimage.2016.10.034. Epub 2016 Oct 22. PMID 27780778
- [Result] Gorka AX, Torrisi S, Shackman AJ, Grillon C, Ernst M. Intrinsic functional connectivity of the central nucleus of the amygdala and bed nucleus of the stria terminalis. Neuroimage. 2018 Mar;168:392-402. doi: 10.1016/j.neuroimage.2017.03.007. Epub 2017 Apr 6. PMID 28392491
- [Result] Cornwell BR, Garrido MI, Overstreet C, Pine DS, Grillon C. The Unpredictive Brain Under Threat: A Neurocomputational Account of Anxious Hypervigilance. Biol Psychiatry. 2017 Sep 15;82(6):447-454. doi: 10.1016/j.biopsych.2017.06.031. Epub 2017 Jul 6. PMID 28838469
- [Result] Torrisi S, Chen G, Glen D, Bandettini PA, Baker CI, Reynolds R, Yen-Ting Liu J, Leshin J, Balderston N, Grillon C, Ernst M. Statistical power comparisons at 3T and 7T with a GO / NOGO task. Neuroimage. 2018 Jul 15;175:100-110. doi: 10.1016/j.neuroimage.2018.03.071. Epub 2018 Apr 3. PMID 29621615
- [Derived] Philips RT, Torrisi SJ, Gorka AX, Grillon C, Ernst M. Dynamic Time Warping Identifies Functionally Distinct fMRI Resting State Cortical Networks Specific to VTA and SNc: A Proof of Concept. Cereb Cortex. 2022 Mar 4;32(6):1142-1151. doi: 10.1093/cercor/bhab273. PMID 34448816
- [Derived] Balderston NL, Flook E, Hsiung A, Liu J, Thongarong A, Stahl S, Makhoul W, Sheline Y, Ernst M, Grillon C. Patients with anxiety disorders rely on bilateral dlPFC activation during verbal working memory. Soc Cogn Affect Neurosci. 2020 Dec 24;15(12):1288-1298. doi: 10.1093/scan/nsaa146. PMID 33150947
- [Derived] Robinson OJ, Pike AC, Cornwell B, Grillon C. The translational neural circuitry of anxiety. J Neurol Neurosurg Psychiatry. 2019 Dec;90(12):1353-1360. doi: 10.1136/jnnp-2019-321400. Epub 2019 Jun 29. PMID 31256001
- [Derived] Gorka AX, Fuchs B, Grillon C, Ernst M. Impact of induced anxiety on neural responses to monetary incentives. Soc Cogn Affect Neurosci. 2018 Nov 8;13(11):1111-1119. doi: 10.1093/scan/nsy082. PMID 30289497
- [Derived] Torrisi S, Gorka AX, Gonzalez-Castillo J, O'Connell K, Balderston N, Grillon C, Ernst M. Extended amygdala connectivity changes during sustained shock anticipation. Transl Psychiatry. 2018 Jan 31;8(1):33. doi: 10.1038/s41398-017-0074-6. PMID 29382815
- [Derived] Balderston NL, Liu J, Roberson-Nay R, Ernst M, Grillon C. The relationship between dlPFC activity during unpredictable threat and CO2-induced panic symptoms. Transl Psychiatry. 2017 Nov 30;7(12):1266. doi: 10.1038/s41398-017-0006-5. PMID 29213110
- [Derived] Balderston NL, Hsiung A, Ernst M, Grillon C. Effect of Threat on Right dlPFC Activity during Behavioral Pattern Separation. J Neurosci. 2017 Sep 20;37(38):9160-9171. doi: 10.1523/JNEUROSCI.0717-17.2017. Epub 2017 Aug 21. PMID 28842415
- [Derived] Balderston NL, Hale E, Hsiung A, Torrisi S, Holroyd T, Carver FW, Coppola R, Ernst M, Grillon C. Threat of shock increases excitability and connectivity of the intraparietal sulcus. Elife. 2017 May 30;6:e23608. doi: 10.7554/eLife.23608. PMID 28555565
- [Derived] Torrisi S, Robinson O, O'Connell K, Davis A, Balderston N, Ernst M, Grillon C. The neural basis of improved cognitive performance by threat of shock. Soc Cogn Affect Neurosci. 2016 Nov;11(11):1677-1686. doi: 10.1093/scan/nsw088. Epub 2016 Jun 30. PMID 27369069
- [Derived] Balderston NL, Vytal KE, O'Connell K, Torrisi S, Letkiewicz A, Ernst M, Grillon C. Anxiety Patients Show Reduced Working Memory Related dlPFC Activation During Safety and Threat. Depress Anxiety. 2017 Jan;34(1):25-36. doi: 10.1002/da.22518. Epub 2016 Apr 25. PMID 27110997
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-M-0321.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 participants were screen failure and two participants withdrew prior to start of study.
Pre-assignment Details: Participants had the option to volunteer for one or more sub-study
Groups:
- Healthy Volunteers: Healthy volunteers participated in one or more sub-studies: Perception, Memory, Resting State, Passive Presentation, Loss Aversion Task, Motivation/reward, valence/salience study (ValSal Task)) and underwent Functional magnetic resonance imaging (fMRI) and/or magneto-encephalography (MEG).
- Patients: Participants with diagnosis of generalized anxiety disorder (GAD), panic disorder, social anxiety disorder (SAD), specific phobia, posttraumatic stress disorder (PTSD), or major depression participated in one or more sub-studies: Perception, Memory, Resting State, Passive Presentation, Loss Aversion Task, Motivation/reward, valence/salience study (ValSal Task)) and underwent Functional magnetic resonance imaging (fMRI).
Period: Overall Study Participants
Arm/Group | Healthy Volunteers | Patients
Started | 921 | 142
Completed | 921 | 142
Not Completed | 0 | 0
Period: Perception Study
Arm/Group | Healthy Volunteers | Patients
Started | 396 | 4
Completed | 396 | 4
Not Completed | 0 | 0
Period: Memory Study
Arm/Group | Healthy Volunteers | Patients
Started | 165 (Include 68 participants who also completed the perception study) | 50
Completed | 165 | 50
Not Completed | 0 | 0
Period: Resting State Study
Arm/Group | Healthy Volunteers | Patients
Started | 218 (Include 19 participants from the perception study and nine participants from the memory study) | 57 (Include one participant from the perception study and three participants from the memory study)
Completed | 218 | 57
Not Completed | 0 | 0
Period: Passive Presentation Study
Arm/Group | Healthy Volunteers | Patients
Started | 57 (Include 16 participants from the perception study, 29 participants from the memory study, and eight participants from the resting state study) | 0
Completed | 57 | 0
Not Completed | 0 | 0
Period: Loss Aversion Task
Arm/Group | Healthy Volunteers | Patients
Started | 14 (Include one participant from the perception study, two participants from the memory study, and seven participants from the resting state study) | 22 (Include 13 participants from the resting state study)
Completed | 14 | 22
Not Completed | 0 | 0
Period: Motivation Task
Arm/Group | Healthy Volunteers | Patients
Started | 264 (Include 14 participants from the perception study, three participants from the memory study, 57 participants from the resting state study, and three participants from the loss aversion task) | 37 (Include one participant from the perception study, 17 participants from the resting state study, and nine participants from the loss aversion task)
Completed | 264 | 37
Not Completed | 0 | 0
Period: Valence/Salience Study (ValSal Task)
Arm/Group | Healthy Volunteers | Patients
Started | 118 (Include seven participants from the perception study, one participant from the memory study, 66 participants from the resting state study, two participants from the loss aversion study, and six participants from the motivation task) | 32 (Include one participant from the perception study, 12 participants from the resting state study, one participant from the loss aversion study, and two participants from the motivation task)
Completed | 118 | 32
Not Completed | 0 | 0
Period: Active Avoidance and Sustained Attention
Arm/Group | Healthy Volunteers | Patients
Started | 162 (Include 38 participants from the perception study, 33 participants from the memory study, 73 participants from the resting state study, two participants from the passive presentation study, two participants from the loss aversion study, and seven participants from the motivation task) | 58 (Include one participant from the perception study, 19 participants from the memory study, 30 participants from the resting state study, six participants from the loss aversion study, one participant from the motivation task, and one participant from the valence/salience study)
Completed | 162 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Perception Study: Participants identified the expression on faces or identified the emotion of a word and were asked to respond during these stimuli themselves and during neutral pictures which were paired with these stimuli. Participants could also be asked to judge how long stimuli remained on the screen by making a button press denoting the relative duration of these stimuli compared to durations they learned.
- Memory Study: Participants performed one or more memory tasks: a) navigated a virtual reality water maze with a joystick to learn the location of an escape platform; b) Behavioral Pattern Separation (BPS) task which consisted of two phases - first participants assign an indoor/outdoor verdict to pictures of neutral objects and completed a memory test. Lastly, participants were asked to remember verbal and nonverbal stimuli which consisted of words, pictures, letters or spatial locations in series of stimuli.
- Resting State Study: Participants laid still with their eyes open and stared at a fixation cross for 6-9 minutes without falling asleep. During a resting state run, participants did not engage in any task. However, on some rest runs, they were under the threat of a shock or safe from shock.
- Passive Presentation Study: Participants engaged in simple, passive experience (visual, auditory, tactile) to measure sensory responses under threat and safe conditions. Participants were asked to remain attentive to whether they were at risk of receiving shock or safe from shocks but did not need to respond to the stimuli.
- Loss Aversion Task: Participants decided between taking or dismissing a series of monetary gambles.
- Motivation Task (Monetary Incentive Delay (MID) Subjects): Participants performed one of two versions of the MID task. The first version of the task examined the effect of threat of shock on goal driven/motivational stimuli where subjects made speeded responses to a central target under conditions of potential monetary gain, loss, or neutrality during threat of shock and during safety. During the second version, participants performed the MID task within the MRI scanner.
- Valence/Salience Study (ValSal Task): Participants completed the ValSal task involving two motivated behaviors, valence and salience. Valence compared the positive versus negative values tagged to stimuli/situations. Salience examined the subjective importance of stimuli/situations.
- Active Avoidance and Sustained Attention Tasks: In the active avoidance signal task (AAST), participants performed a modified version of the threat paradigm during which, they held down a button and view sequentially presented pairs of colored squares and were instructed to lift their finger when they see the medium-medium color combination (i.e. "go" trials), and to refrain from lifting their finger during all other combinations (i.e. "stop" trials). Participants performed alternating blocks in safe and threat conditions, and each block consisted of a series of "go" and "stop" trials.
  In the sustained attention to response task (SART), subjects participated in go/nogo during periods of threat of shocks and periods of safety, when no shock could be administered.
- Total: Total of all reporting groups
Arm/Group | Perception Study | Memory Study | Resting State Study | Passive Presentation Study | Loss Aversion Task | Motivation Task (Monetary Incentive Delay (MID) Subjects) | Valence/Salience Study (ValSal Task) | Active Avoidance and Sustained Attention Tasks | Total
Number analyzed (Participants) | 400 | 147 | 243 | 4 | 13 | 197 | 52 | 7 | 1063
Age, Categorical [Count of Participants; unit: Participants] — Population: Analysis is a breakout of the two groups in the study
  Participants
    Healthy Volunteers: number analyzed (Participants) | 396 | 97 | 190 | 4 | 4 | 187 | 36 | 7 | 921
    Healthy Volunteers: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Healthy Volunteers: Between 18 and 65 years | 396 | 97 | 190 | 4 | 4 | 187 | 36 | 7 | 921
    Healthy Volunteers: >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patients: number analyzed (Participants) | 4 | 50 | 53 | 0 | 9 | 10 | 16 | 0 | 142
    Patients: <=18 years | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0
    Patients: Between 18 and 65 years | 4 | 50 | 53 |  | 9 | 10 | 16 | 0 | 142
    Patients: >=65 years | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analysis is a breakout of the two groups in the study
  Participants
    Healthy Volunteers: number analyzed (Participants) | 396 | 97 | 190 | 4 | 4 | 187 | 36 | 7 | 921
    Healthy Volunteers: Female | 201 | 48 | 106 | 1 | 3 | 83 | 21 | 3 | 466
    Healthy Volunteers: Male | 195 | 49 | 84 | 3 | 1 | 104 | 15 | 4 | 455
    Patients: number analyzed (Participants) | 4 | 50 | 53 | 0 | 9 | 10 | 16 | 0 | 142
    Patients: Female | 2 | 33 | 41 | 0 | 9 | 9 | 10 | 0 | 104
    Patients: Male | 2 | 17 | 12 | 0 | 0 | 1 | 6 | 0 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Analysis is a breakout of the two groups in the study
  Participants
    Healthy Volunteers: number analyzed (Participants) | 396 | 97 | 190 | 4 | 4 | 187 | 36 | 7 | 921
    Healthy Volunteers: Hispanic or Latino | 21 | 5 | 21 | 0 | 1 | 15 | 4 | 0 | 67
    Healthy Volunteers: Not Hispanic or Latino | 367 | 92 | 167 | 4 | 3 | 165 | 32 | 7 | 837
    Healthy Volunteers: Unknown or Not Reported | 8 | 0 | 2 | 0 | 0 | 7 | 0 | 0 | 17
    Patients: number analyzed (Participants) | 4 | 50 | 53 | 0 | 9 | 10 | 16 | 0 | 142
    Patients: Hispanic or Latino | 0 | 4 | 7 | 0 | 0 | 1 | 1 | 0 | 13
    Patients: Not Hispanic or Latino | 4 | 44 | 44 | 0 | 9 | 9 | 15 | 0 | 125
    Patients: Unknown or Not Reported | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Analysis is a breakout of the two groups in the study
  Participants
    Healthy Volunteers: number analyzed (Participants) | 396 | 97 | 190 | 4 | 4 | 187 | 36 | 7 | 921
    Healthy Volunteers: American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Healthy Volunteers: Asian | 47 | 20 | 40 | 0 | 1 | 15 | 12 | 0 | 135
    Healthy Volunteers: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
    Healthy Volunteers: Black or African American | 80 | 26 | 47 | 0 | 0 | 42 | 6 | 2 | 203
    Healthy Volunteers: White | 242 | 45 | 84 | 4 | 2 | 111 | 17 | 4 | 509
    Healthy Volunteers: More than one race | 8 | 2 | 8 | 0 | 0 | 4 | 1 | 1 | 24
    Healthy Volunteers: Unknown or Not Reported | 19 | 2 | 10 | 0 | 1 | 15 | 0 | 0 | 47
    Patients: number analyzed (Participants) | 4 | 50 | 53 | 0 | 9 | 10 | 16 | 0 | 142
    Patients: American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Patients: Asian | 0 | 2 | 5 | 0 | 3 | 1 | 1 | 0 | 12
    Patients: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patients: Black or African American | 2 | 11 | 10 | 0 | 1 | 1 | 4 | 0 | 29
    Patients: White | 2 | 28 | 30 | 0 | 4 | 8 | 9 | 0 | 81
    Patients: More than one race | 0 | 7 | 4 | 0 | 0 | 0 | 2 | 0 | 13
    Patients: Unknown or Not Reported | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Average Correlations Between Average Time Series - Left & Right Hemisphere of the Brain
Description: The average bed nucleus of the stria terminalis (BNST) correlations between all averaged time series were extracted from the raters' individual masks. Blood Oxygenation Level Dependent (BOLD) signals were used to extract a mean time series from the BNST masks. This time series was correlated across the rest of the brain using 3dTcorr1D, which computes the correlation coefficient between each voxel time series. Raters were blinded to subject identity for subjective sensory effects at high field and inter-rater and volume measurements for the drawn BNST masks. Correlations were calculated between average time series extracted between all raters' masks for each subject. Two separate analyses for the left and right BNSTs were performed.
Time Frame: 10 minutes
Population: Analysis was done on a sample of healthy participants
Measure: Mean (Standard Deviation); unit: correlation coefficient (r)
Groups:
- Healthy Volunteers: Healthy volunteers underwent Functional magnetic resonance imaging (fMRI) and/or magneto-encephalography (MEG).
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 27
correlation coefficient (r)
  Left BNST | 0.9 (0.08)
  Right BNST | 0.92 (0.07)
Statistical Analysis 1: Comparison: Healthy Volunteers; Test type: Other; p < 0.001, ANOVA

2. Primary Outcome: Difference in Volume - Left & Right Habenula
Description: Images were acquired on a 7 T Siemens Magnetom MRI with a 32-channel head coil over 10 minutes. Participants were instructed to keep their eyes open and look at a white fixation cross on a black background during image acquisition. Following manual tracing of the habenula, the volumes of the left and right habenulae for each subject were computed separately. The left and right habenula volumes were then compared using a paired t-test.
Time Frame: 10 minutes
Population: Analysis was done on a pilot sample of healthy volunteer participants
Measure: Mean (Standard Deviation); unit: mm^3
Groups:
- Healthy Volunteer: Healthy volunteers underwent Functional magnetic resonance imaging (fMRI) and/or magneto-encephalography (MEG).
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 32
mm^3
  Left Habenula | 18.8 (6)
  Right Habenula | 14.9 (4)
Statistical Analysis 1: Comparison: Healthy Volunteer; Test type: Other; p = 0.000093, t-test, 2 sided

3. Primary Outcome: Percent of Correct No Button Presses During Functional MRI
Description: Subjects participated in go/nogo (91% GO trials with the " = " symbol indicating button push and 9% NOGO trials with the "O" symbol indicating no push)) task condition during 3 Tesla (3T) or 7 Tesla (7T) functional MRI with periods of threat of shocks and periods of safety when no shock could be administered. During the GNG stimuli were presented on a monitor and randomly distributed. A correct go hit was a response recorded during these 2000 ms to a go trial. Similarly, a correct nogo omission was a no response during the same period to a nogo trial. Performance was first averaged across condition (threat, safe) and trial type (go, nogo) by dividing the number of correct responses by the total number of each trial type. The NOGO and GO behavioral effects were then separately compared between 3T and 7T strength. Accuracy was measured as a percent of correct button presses during fMRI (3T or 7T).
Time Frame: 2000 milliseconds during trial
Population: Analysis included only participants who completed the Sustained Attention to Response Task (SART)
Measure: Mean (Standard Deviation); unit: Percentage of accurate responses
Groups:
- Healthy Volunteers - 3T fMRI: Healthy volunteers underwent 3T Functional magnetic resonance imaging (fMRI) and participated in go/nogo trial under threat of shock or no shock
- Healthy Volunteers - 7T fMRI: Healthy volunteers underwent 7T Functional magnetic resonance imaging (fMRI) and participated in go/nogo trial under threat of shock or no shock
Arm/Group | Healthy Volunteers - 3T fMRI | Healthy Volunteers - 7T fMRI
Number analyzed (Participants) | 31 | 31
Percentage of accurate responses
  NOGO Trials | 71 (20) | 76 (15)
  GO Trials | 99 (3) | 95 (7)

ADVERSE EVENTS:
Time Frame: Up to three hours in a single day visit for a maximum of three visits
Groups:
- Perception Study - Healthy Volunteer; Perception Study - Patient: Participants identified the expression on faces or identified the emotion of a word and were asked to respond during these stimuli themselves and during neutral pictures which were paired with these stimuli. Participants could also be asked to judge how long stimuli remained on the screen by making a button press denoting the relative duration of these stimuli compared to durations they learned.
- Memory Study - Healthy Volunteer; Memory Study - Patient: Participants performed one or more memory tasks: a) navigated a virtual reality water maze with a joystick to learn the location of an escape platform; b) Behavioral Pattern Separation (BPS) task which consisted of two phases - first participants assign an indoor/outdoor verdict to pictures of neutral objects and completed a memory test. Lastly, participants were asked to remember verbal and nonverbal stimuli which consisted of words, pictures, letters or spatial locations in series of stimuli.
- Resting State Study - Healthy Volunteer; Resting State Study - Patient: Participants laid still with their eyes open and stared at a fixation cross for 6-9 minutes without falling asleep. During a resting state run, participants did not engage in any task. However, on some rest runs, they were under the threat of a shock or safe from shock.
- Passive Presentation Study - Healthy Volunteer: Participants engaged in simple, passive experience (visual, auditory, tactile) to measure sensory responses under threat and safe conditions. Participants were asked to remain attentive to whether they were at risk of receiving shock or safe from shocks but did not need to respond to the stimuli.
- Loss Aversion Task - Healthy Volunteer; Loss Aversion Task - Patient: Participants decided between taking or dismissing a series of monetary gambles.
- Motivation Task (Monetary Incentive Delay (MID) Study) - Healthy Volunteer; Motivation Task (Monetary Incentive Delay (MID) Study) - Patient: Participants performed one of two versions of the MID task. The first version of the task examined the effect of threat of shock on goal driven/motivational stimuli where subjects made speeded responses to a central target under conditions of potential monetary gain, loss, or neutrality during threat of shock and during safety. During the second version, participants performed the MID task within the MRI scanner.
- Valence/Salience Study (ValSal Task) - Healthy Volunteer; Valence/Salience Study (ValSal Task) - Patient: Participants completed the ValSal task involving two motivated behaviors, valence and salience. Valence compared the positive versus negative values tagged to stimuli/situations. Salience examined the subjective importance of stimuli/situations.
- Active Avoidance and Sustained Attention Tasks - Healthy Volunteer; Active Avoidance and Sustained Attention Tasks - Patient: In the active avoidance signal task (AAST), participants performed a modified version of the threat paradigm during which, they held down a button and view sequentially presented pairs of colored squares and were instructed to lift their finger when they see the medium-medium color combination (i.e. "go" trials), and to refrain from lifting their finger during all other combinations (i.e. "stop" trials). Participants performed alternating blocks in safe and threat conditions, and each block consisted of a series of "go" and "stop" trials.
  In the sustained attention to response task (SART), subjects participated in go/nogo during periods of threat of shocks and periods of safety, when no shock could be administered.
Arm/Group | Perception Study - Healthy Volunteer | Perception Study - Patient | Memory Study - Healthy Volunteer | Memory Study - Patient | Resting State Study - Healthy Volunteer | Resting State Study - Patient | Passive Presentation Study - Healthy Volunteer | Loss Aversion Task - Healthy Volunteer | Loss Aversion Task - Patient | Motivation Task (Monetary Incentive Delay (MID) Study) - Healthy Volunteer | Motivation Task (Monetary Incentive Delay (MID) Study) - Patient | Valence/Salience Study (ValSal Task) - Healthy Volunteer | Valence/Salience Study (ValSal Task) - Patient | Active Avoidance and Sustained Attention Tasks - Healthy Volunteer | Active Avoidance and Sustained Attention Tasks - Patient
All-Cause Mortality (participants affected / at risk) | 0/396 | 0/4 | 0/165 | 0/50 | 0/218 | 0/57 | 0/57 | 0/14 | 0/22 | 0/264 | 0/37 | 0/118 | 0/32 | 0/162 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/396 | 0/4 | 0/165 | 0/50 | 0/218 | 0/57 | 0/57 | 0/14 | 0/22 | 0/264 | 0/37 | 0/118 | 0/32 | 0/162 | 0/58
Other Adverse Events (participants affected / at risk) | 0/396 | 0/4 | 0/165 | 0/50 | 0/218 | 0/57 | 0/57 | 0/14 | 0/22 | 0/264 | 0/37 | 0/118 | 0/32 | 0/162 | 0/58

LIMITATIONS AND CAVEATS:
This protocol was a series of sub-studies using sample subjects which explains the number of participants per study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT00047853/Prot_SAP_000.pdf